CLINICAL TRIAL: NCT01449617
Title: Observational Study on Predictive Value for Vascular Events of Residual Platelet Aggregation in Patients on Antiplatelet Therapy After Carotid Angioplasty With Stenting
Brief Title: Residual Platelet Reactivity in Patients on Antiplatelet Therapy After Carotid Angioplasty With Stenting
Acronym: ARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Perugia (Other)
Collaborators: University Of Perugia (Other)
Responsible Party: Principal Investigator, Paolo Gresele, Clinical Investigator, Azienda Ospedaliera di Perugia
Other Study IDs: UniPG; CEAS (Other: Comitato Etico delle Aziende Sanitarie dell'Umbria)
Record Dates: First submitted 2011-06-23; First posted 2011-10-10 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Carotid Artery Disease
Keywords: Carotid stenosis; Aspirin plus Clopidogrel; Residual platelet reactivity
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples, plasma samples, serum samples, urines.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aspirin plus clopidogrel: Patients undergoing stenting for critical carotid stenosis, either symptomatic (previous events of cerebral ischemia) or asymptomatic, undergoing CAS.
  Interventions: Drug: Aspirin plus clopidogrel

INTERVENTIONS:
Drug: Aspirin plus clopidogrel — Clopidogrel, will be started 48 hours before the procedure with a loading dose of of 300mg and continued at 75mg/day.
  Aspirin will be given at the dose of 100-325mg/day.
  Other Names: Cardioaspirina; Plavix

SUMMARY:
A carotid stenosis is treated with invasive procedures of revascularization when the lumen is reduced by more than 70% or when the lumen is reduced by more than 50% in patients who have had symptoms attributable to the affected carotid district in last the 6 months.

Two options for the treatment of patients with carotid stenosis exist currently: the traditional surgical intervention of removal of the plaque by carotid endoarterectomy (CEA)and percutaneous transluminal carotid angioplasty with a balloon associated to the positioning of a stent through a catheter brought directly in the carotid artery (CAS).

The main complication of both the procedures is early thrombosis, a phenomenon in which platelets play a central role. The importance of an effective inhibition of platelet activation in these patients has been widely demonstrated.

Clinical studies in patients undergoing PTCA have demonstrated that the optimal treatment for the prevention of stent thrombosis is a dual antiplatelet regimen with aspirin plus clopidogrel, as compared with the single drugs. Given that no specific clinical trial has assessed the best antiplatelet therapeutic regimen in CAS with stenting, by extension from these findings in ischemic heart disease CAS patients are treated with aspirin plus clopidogrel.

Several studies have demonstrated that an elevated residual platelet reactivity despite treatment with clopidogrel is associated to an increased risk of major adverse cardiovascular events (MACE) after stenting for coronary disease.

No data are instead available on the possible predictive value of residual platelet reactivity for the incidence of ischemic cardiovascular events in patients with atherosclerotic carotid disease undergoing CAS with stenting.

Aim of the study will be to assess the predictive value of residual platelet reactivity, as measured by different laboratory tests in patients undergoing CAS with stenting and treated with aspirin plus clopidogrel, for the incidence of cardiovascular complications (major adverse ischemic events).

DETAILED DESCRIPTION:
STUDY DESIGN The study will enroll 110 patients undergoing stenting for critical carotid stenosis, either symptomatic (previous events of cerebral ischemia) or asymptomatic, undergoing CAS.

All patients undergoing CAS in our Center and that fit the predefined Criteria will be enrolled in the study. Dual-antiplatelet treatment with aspirin and clopidogrel will be administered to all patients with the same modalities in use for coronary heart disease patients undergoing PTCA.

Implanted stents after CAS will be in all patients bare metal stents (BMS) and therefore, by analogy with the studies in ACS, the duration of dual-antiplatelet treatment will be of one month; later all patients will be continued indefinitely on aspirin.

Clopidogrel, will be started 48 hours before the procedure with a loading dose of of 300mg and continued at 75mg/day; aspirin will be given at the dose of 100-325mg/day.

Platelet reactivity assessment will be carried-out:

* before intervention,
* after 1 week of treatment,
* after 1 month of treatment
* after 1 year. All patients will be recalled for clinical examination at 1 and 6 months and at 1 year.

ELIGIBILITY:
Inclusion criteria

* Informed written consent
* No contraindications to dual-antiplatelet treatment

Exclusion criteria

* Age < 18 or > 80 years old
* Use of oral anticoagulants
* Use of dipyridamole, cilostazol, NSAIDs
* Myeloproliferative syndrome or paraproteinemia
* Liver or kidney failure
* Thrombocytopathies
* Platelets count < 100000 or > 450000/µl
* Haemoglobin < 8g/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 506 patients undergoing stenting for critical carotid stenosis, either symptomatic (previous events of cerebral ischemia) or asymptomatic, undergoing CAS.
Sampling Method: Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2010-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in Platelet reactivity | 1, 6 and 12 months
  assessed by VerifyNow (ASA and P2Y12 cartridges), Multiplate (ASA and ADP cartridges), PFA100 (coll/epi; coll/adp; coll/P2Y12 cartridges)
Change in Occurrence of stroke | 1, 6 and 12 months
  assessed by subsequent follow-up
Change in Occurence of myocardial infarction | 1, 6 and 12 months
  assessed by subsequent follow-up
Change in occurrence of lower limb ischemia | 1, 6 and 12 months
  assessed by subsequent follow-up

SECONDARY OUTCOMES:
Change in Incidence of restenosis | 6 and 12 months
  assessed by Eco Color Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gresele, Prof., Principal Investigator — University Of Perugia
Locations (1):
- Azienda Ospedaliera di Perugia, Perugia, Italy, Italy